CLINICAL TRIAL: NCT04830709
Title: Prospective Non-interventional Study to Collect Real-world Clinical and Patient-reported Outcome Data in Ovarian Cancer Patients Eligible for First-line Platinum-based Chemotherapy and Intended for BRCA/HRD Testing
Brief Title: Non-interventional Study to Collect Real-world Clinical and Patient-reported Outcomes in Ovarian Cancer
Acronym: SCOUT-1
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: North-Eastern German Society of Gynecological Oncology e.V. (NOGGO e.V.) (Unknown)
Responsible Party: Sponsor
Other Study IDs: D0817R00030
Record Dates: First submitted 2021-03-18; First posted 2021-04-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
Keywords: Patient reported outcome (PRO),; advanced Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PARPi maintenance cohort (PMC): patients who received at least one dose of PARPi as 1L MTX after 1L platinum-based CTX
- Bevacizumab maintenance cohort (BMC): patients who continue to receive at least one dose of bevacizumab after 1L platinum-based CTX and who have not received PARPi MTX treatment
- No maintenance cohort (NMC): patients who never received any 1L MTX treatment (PARPi or bevacizumab)

SUMMARY:
This prospective non-interventional study is intended to generate new data and insights into first-line (1L) treatment of newly diagnosed advanced high-grade epithelial Ovarian cancer (OC) in Germany relevant for patients, physicians and payers. It will capture the influence of 1L Poly ADP ribose polymerase inhibitor (PARPi) maintenance treatment (MTX) on medical routine in Germany, especially on:

* outcome of the 3-steps 1L treatment phase (including surgery, Chemotherapy (CTX) and MTX) including the potential of patients with primary advanced OC to be cured,
* patient's follow-up (FU) during and after MTX therapy,
* patient-reported outcomes (PROs), experiences and needs,
* physician's experience,
* BRCA/HRD and genomic scar testing behavior at diagnosis/during 1L therapy,
* patient selection for different 1L systemic treatment approaches,
* use and safety of drugs,
* treatment sequence in case of recurrence

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Women aged ≥ 18 years
3. Newly diagnosed with primary advanced (FIGO stages III and IV) high-grade epithelial ovarian cancer (including fallopian tube and/or primary peritoneal cancer)
4. For patients who qualify for primary debulking surgery, all surgical procedures must be completed prior to enrollment
5. BRCA mutation test (routinely analyzed germline and/or somatic BRCA1/2 status alone or as part of HRD status determination) already performed or initiated/intended
6. First-line platinum-based chemotherapy planned or a maximum of 3 cycles already received with no sign of disease progression. Total number of cycles after enrollment should be decided individually for each single patient by the treating physician. In case of neoadjuvant chemotherapy and interval debulking surgery, the patient should be enrolled after completion of surgical procedure and at the time of the 1st post-surgery cycle of platinum-based chemotherapy.
7. Willing and able to report PROs electronically
8. Women of childbearing potential must use two forms of reliable contraception according to standard of care

Exclusion Criteria:

1. Pregnancy or breast-feeding 2. Current or planned participation in an interventional clinical trial on first-line treatment of OC 3. Current or upcoming systemic treatment of any tumor other than OC 4. Not eligible for platinum-based chemotherapy or early progress during the cycles of first-line platinum-based chemotherapy prior to enrollment

-

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approx. 750 patients with newly diagnosed advanced (FIGO stage III or IV) high-grade epithelial ovarian, fallopian-tube, or primary peritoneal cancer are planned to be included in the study in a consecutive manner
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2033-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | date of 1st dose of 1L platinum-based CTX to disease progression (investigator-assessed according to clinical routine) or death of any cause, whichever came first, assessed up to 84 months
  The primary outcome is progression-free survival (PFS) defined as time from 1st dose of 1L platinum-based CTX to disease progression (investigator-assessed according to clinical routine) or death of any cause. Methods and intervals for tumor assessments are at the discretion of the treating physician. Details on progression incl. the procedure used to confirm progression (e.g. symptoms, ultrasound, x-ray, CT, MRI) will be captured in the eCRF.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | time of 1st dose of 1L platinum-based CTX to disease progression (investigator-assessed according to clinical routine) or death of any cause, whichever came first, assessed up to 84 months
  Recurrence-free survival (RFS) is time from 1st dose of 1L platinum-based CTX to disease recurrence (investigator-assessed according to clinical routine) or death of any cause defined as in patients with no evidence of disease (NED) following platinum-based CTX
Progression-/recurrence-free survival rate | percentage of patients without disease progression/recurrence alive at 2, 3, 5 and 7 years
  Progression-/recurrence-free survival rate is defined as the percentage of patients without disease progression/recurrence alive at 2, 3, 5 and 7 years derived by Kaplan-Meier methods in the full analysis set/subset of patients with NED; Patients within NED subset will be considered as long-term disease-free survivors (potentially cured) if they are disease free for the whole period of 7 years
Time to first subsequent therapy (TFST) | time from 1st dose of 1L platinum-based CTX to the 1st dose of subsequent therapy or death of any cause, whichever came first, assessed up to 84 months
  Time to first subsequent therapy (TFST) is defined as time from 1st dose of 1L platinum-based CTX to the 1st dose of subsequent therapy or death of any cause;
Second progression-free survival (PFS2) | time from 1st dose of 1L platinum-based CTX to second disease progression (investigator-assessed according to clinical routine) or death of any cause, whichever came first, assessed up to 84 months
  Second progression-free survival (PFS2) is defined as time from 1st dose of 1L platinum-based CTX to second disease progression (investigator-assessed according to clinical routine) or death of any cause. Methods and intervals of tumor assessments are at the discretion of the treating physician and will be recorded in the eCRF
Time to second subsequent therapy (TSST) | time from 1st dose of 1L platinum-based CTX to the 1st dose of second subsequent therapy or death of any cause, whichever came first, assessed up to 84 months
  Time to second subsequent therapy (TSST) as time from 1st dose of 1L platinum-based CTX to the 1st dose of second subsequent therapy or death of any cause
3rd, 4th, 5th ff. progression-free survival (PFSx = PFS3, 4, 5 ff.) | time from 1st dose of 1L platinum-based CTX to 3rd, 4th, 5th and later disease progression [investigator-assessed according to clinical routine] or death of any cause, whichever came first, assessed up to 84 months
  3rd, 4th, 5th ff. progression-free survival (PFSx = PFS3, 4, 5 ff.) is defined as time from 1st dose of 1L platinum-based CTX to 3rd, 4th, 5th and later disease progression [investigator-assessed according to clinical routine] or death of any cause). Methods and intervals of tumor assessments are at the discretion of the treating physician and will be recorded in the eCRF
Time to 3rd, 4th, 5th and later subsequent therapy (TST 3rd, 4th, 5th ff.) | defined as time from 1st dose of 1L platinum-based CTX to the 1st dose of 3rd, 4th, 5th and later subsequent therapy or death of any cause, whichever came first, assessed up to 84 months
  Time to 3rd, 4th, 5th and later subsequent therapy (TST 3rd, 4th, 5th ff.) is defined as time from 1st dose of 1L platinum-based CTX to the 1st dose of 3rd, 4th, 5th and later subsequent therapy or death of any cause
Overall survival (OS) | time from 1st dose of 1L platinum-based CTX to death of any cause, assessed up to 84 months
  Overall survival (OS) is defined as time from 1st dose of 1L platinum-based CTX to death of any cause
Patient-reported health-related quality of life (HRQoL) - EQ-5D questionnaire | during observation period of the study: primary therapy/maintenance, recurrence/progression, subsequent treatments, up to 84 months
  The EQ-5D is a standardized measure of health status applicable to a wide range of health conditions and treatments designed by the EuroQoL Group (EQ). It consists of the EQ-5D descriptive system, which comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with each dimension having 5 levels (5L), and the EQ visual analogue scale (EQ VAS).
Patient-reported health-related quality of life (HRQoL) - FACT-O questionnaire | during observation period of the study: primary therapy/maintenance, recurrence/progression, subsequent treatments, up to 84 months
  Functional Assessment of Cancer Therapy-Ovarian Cancer (FACT-O) Quality of life of women with OC is assessed by means of the FACT-O questionnaire. It contains questions addressing the most frequent problems of cancer patients: physical well-being, social/family well-being, emotional well-being, functional well-being, as well as additional concerns specific to OC (such as female-specific concerns and abdominal problems)
Patient-reported health-related quality of life (HRQoL) - MOSTv2 questionnaire | during observation period of the study: primary therapy/maintenance, recurrence/progression, subsequent treatments, up to 84 months
  Measure of Ovarian Symptoms and Treatment concerns Version 2 (MOSTv2) The MOST quantifies patient-reported symptom burden, adverse effects, and symptom benefit in OC patients. MOSTv2 has 24 items and five multi-item scales: abdominal symptoms (MOST-Abdo), disease or treatment-related symptoms (MOST-DorT), chemotherapy-related symptoms (MOST-Chemo), psychological symptoms (MOST-Psych), and MOST-Well-being
Patient-reported health-related quality of life (HRQoL) - PGI-S questionnaire | during observation period of the study: primary therapy/maintenance, recurrence/progression, subsequent treatments, up to 84 months
  Patient global impression of severity of cancer symptoms (PGI-S) is a one-item scale to assess a patient's impression of disease severity on a four-point scale from normal to severe.

OTHER OUTCOMES:
Patient's expectations/needs | at baseline, once a year during routine visits, up to 84 months
  Patient's expectations/needs for support/information/education regarding the disease itself and the current therapy (systemic therapies during surgery, CTX, MTX, FU, long-term survivor) as determined by unstandardized questionnaire partially based on EXPRESSION IV questionnaire and open questioning
physician's expectations on therapy | at baseline, once a year during routine visits, up to 84 months
  data on the physician's expectations on systemic therapies (unstandardized questionnaire) will be collected after the physician has enrolled the first patient (FPI) and afterwards annually
BRCA mutation testing behavior | documented at baseline
  BRCA mutation testing behavior during clinical routine will be assessed with respect to initiator, time of test initiation, type of sample, variants detected, and turnaround time (TAT: duration from request of the BRCA mutation analysis or receipt of the sample in the laboratory, whichever comes later, and the release of the report). Details will be retrospectively assessed for patients with an already existing test result at study inclusion
HRD testing behavior | documented at baseline
  HRD testing behavior during clinical routine will be assessed with respect to initiator, type of sample, type of test, HRD status result, HRD score, and turnaround time (TAT: duration from request of HRD analysis or receipt of the sample in the laboratory, whichever comes later, and the release of the report). Details will be retrospectively assessed for patients with an already existing test result at study inclusion.
Safety: Collection of Adverse Events (AE) | during routine visits, up to 84 months
  Safety evaluated based on type of Adverse Event (AE), intensity, causal relationship to treatment, duration, handling, outcome, and seriousness
Patient population | at baseline and changes at time points of expected routine visits, up to 84 months
  Patient population described on the basis of:
  * Baseline characteristics
  * Disease history
  * Social status
  * Comorbidities and concomitant treatments

CONTACTS AND LOCATIONS:
Locations (77):
- Germany (77):
  - Research Site, Böblingen, Germany
  - Research Site, Göttingen, Germany
  - Research Site, Nürtingen, Germany
  - Research Site, Osnabrück, Germany
  - Research Site, Rotenburg (Wümme), Germany
  - Research Site, Schwäbisch Hall, Germany
  - Research Site, Aachen
  - Research Site, Amberg
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Baden-Baden
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Borna
  - Research Site, Bottrop
  - Research Site, Brandenburg
  - Research Site, Bremen
  - Research Site, Coburg
  - Research Site, Cologne
  - Research Site, Dessau
  - Research Site, Donauwörth
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Eggenfelden
  - Research Site, Erfurt
  - Research Site, Fürth
  - Research Site, Gelnhausen
  - Research Site, Gera
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanau
  - Research Site, Heilbronn
  - Research Site, Hildesheim
  - Research Site, Homburg
  - Research Site, Itzehoe
  - Research Site, Jena
  - Research Site, Kiel
  - Research Site, Krefeld
  - Research Site, Leipzig
  - Research Site, Limburg
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Mönchengladbach
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Offenburg
  - Research Site, Pforzheim
  - Research Site, Plauen
  - Research Site, Potsdam
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Research Site, Rheine
  - Research Site, Rosenheim
  - Research Site, Rostock
  - Research Site, Saarlouis
  - Research Site, Siegen
  - Research Site, Singen
  - Research Site, Solingen
  - Research Site, Stendal
  - Research Site, Stralsund
  - Research Site, Stuttgart
  - Research Site, Torgau
  - Research Site, Traunstein
  - Research Site, Ulm
  - Research Site, Villingen-Schwenningen
  - Research Site, Wiesbaden
  - Research Site, Winnenden
  - Research Site, Witten
  - Research Site, Wolfsburg
  - Research Site, Worms
  - Research Site, Wuppertal

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home